CLINICAL TRIAL: NCT05118009
Title: Artificial Intelligence Based Rapid Identification of ST-elevation Myocardial Infarction Using Electrocardiogram (ARISE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NDMC2021003
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention will have access to the screening tool.
  Interventions: Other: AI-enabled ECG-based Screening Tool
- Control (No Intervention): Patients randomized to control will continue routine practice.

INTERVENTIONS:
Other: AI-enabled ECG-based Screening Tool — Primary care clinicians in the intervention group had access to the report, which displayed whether the AI-ECG result was positive or negative.The system will send a message to corresponding physicians if positive finding.
  Arms: Intervention

SUMMARY:
This is a randomized controlled trial (RCT) to test a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based supporting tool for improving the diagnosis and management of ST-elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients in emergency department or inpatient department.
* Patients recieved at least 1 ECG examination.

Exclusion Criteria:

* The patients recieved ECG at the period of inactive AI-ECG system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43176 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
E2C (ECG to coronary angiography) time | Within 6 hours
  Time from ECG to activation of coronary angiography for STEMI patients.

SECONDARY OUTCOMES:
E2B (ECG to primary percutaneous coronary intervention) time | Within 6 hours
  Time from ECG to complete of primary percutaneous coronary intervention for STEMI patients.
D2B (Door to Balloon Time) time | Within 6 hours
  Time from first medical contact to complete of primary percutaneous coronary intervention for STEMI patients in emergency department.
D2C (Door to coronary angiography) time | Within 6 hours
  Time from first medical contact to activation of coronary angiography for STEMI patients in emergency department.
Ejection fractrion | Within 3 days
  Ejection fractrion primary percutaneous coronary intervention for STEMI patients.
Highest concentration of high-sensitivity cardiac troponin I | Within 3 days
  After performing an electrocardiogram, the highest concentration of high-sensitivity cardiac troponin I was followed.
Highest concentration of creatine kinase | Within 3 days
  After performing an electrocardiogram, the highest concentration of creatine kinase was followed.
Length of hospitalization | Within 28 days
  After performing an electrocardiogram, the length of hospitalization.
Number of CAG event | Within 6 hours
  Number of CAG event

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No